CLINICAL TRIAL: NCT04701099
Title: Population Pharmacokinetics of Vancomycin, Meropenem, Milrinone, Dexmedetomidine and Fentanyl in Pediatric Patients During Extracorporeal Membrane Oxygenation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-0182
Record Dates: First submitted 2021-01-03; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pediatric Patients Receiving Venoarterial Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At each sampling time, an arterial blood sample (1 to 2 mL) is collected from all subjects during ECMO support and after weaning off ECMO for drug concentration assay (LC-MS/MS, etc.).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On ECMO: patients who is receiving vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl during ECMO support.
- Off ECMO: patients who is receiving vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl after weaning off ECMO.

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) has been used primarily in newborns since it was first successfully implemented in the 1970s, and has recently increased use in infants and young children. Venoarterial ECMO (VA-ECMO) is a temporary mechanical circulatory support for patients with cardiac failure. Because ECMO is invasive, appropriate use of antimicrobial agent, analgesic and sedatives is important to promote recovery. However, a large variability in drugs pharmacokinetics is expected in pediatric ECMO patients due to the combination of ECMO, drug characteristics and disease factor. This study aimed to evaluate whether the PK of drugs is influenced by VA-ECMO and to recommend the optimal dosing strategies for proposed drugs in pediatric patients receiving VA-ECMO.

ELIGIBILITY:
Inclusion Criteria:

* <19 years old
* receiving VA ECMO in Severance Hospital, Yonsei University Health System.
* receiving one of these drugs: vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl
* agreed to participate

Exclusion Criteria:

* receiving drugs that could affect study drug's concentration due to drug-drug interaction

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under the age of 19 who are receiving vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl while using VA ECMO in Severance Hospital, Yonsei University Health System.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-07 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Serum or plasma concentration | Between day0 to day3 during ECMO
  Serum or plasma concentration of vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl
Serum or plasma concentration | Between day0 to day3 after weaning off ECMO
  Serum or plasma concentration of vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl
Pharmacokinetic parameter: Volume of distribution | Between day0 to day3 during ECMO
  Volume of distribution of vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl
Pharmacokinetic parameter: Volume of distribution | Between day0 to day3 after weaning off ECMO
  Volume of distribution of vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl
Pharmacokinetic parameter: Clearance | Between day0 to day3 during ECMO
  Clearance of vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl
Pharmacokinetic parameter: Clearance | Between day0 to day3 after weaning off ECMO
  Clearance of vancomycin or meropenem or milrinone or dexmedetomidine or fentanyl

CONTACTS AND LOCATIONS:
Overall Officials: Yu Rim Shin, Assistant Professor, Principal Investigator — Severance Hospital
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No